CLINICAL TRIAL: NCT07258706
Title: DIVER-TAVI Registry - Demographic and Interpopulation Variations in Evaluation and Results of TAVI
Brief Title: Demographic and Interpopulation Variations in Evaluation and Results of TAVI
Acronym: DIVER-TAVI
Status: Enrolling by invitation | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2025_538
Record Dates: First submitted 2025-09-12; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis; TAVI(Transcatheter Aortic Valve Implantation); Computed Tomography; Inflammatory Response During Cardiac Surgery; Inflammation
Keywords: Aortic stenosis; transcatheter aortic valve implantation; TAVI; Computed Tomography; Inflammation
MeSH Terms: conditions — Aortic Valve Stenosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with aortic stenosis qualified for TAVI: All consecutive patients with severe aortic stenosis qualified for TAVI according to current guidelines
  Interventions: Diagnostic Test: laboratory biomarker analysis; Diagnostic Test: Computed tomography of aortic root and aorta

INTERVENTIONS:
Diagnostic Test: laboratory biomarker analysis — Results of common laboratory tests obtained during routine care in the pre-procedural period (simple blood morphology, creatinine, GFR, NTproBNP). Inflammatory indices - NLR, MLR, PLR
Diagnostic Test: Computed tomography of aortic root and aorta — Results of CT analysis performed as a routine diagnostic examination in the pre-procedural period will be recorded.

SUMMARY:
The aim of the project is to evaluate demographic, clinical, and laboratory variations in patients with aortic stenosis treated with TAVI in different countries. Moreover, the study will evaluate interpopulation differences in aortic root anatomy based on computed tomography analysis.

DETAILED DESCRIPTION:
Aortic stenosis represents the most common valvular heart disease in developed countries, with a significant epidemiologic increase related to the aging population. Currently, surgical and transcatheter interventions are the only therapeutic options, as pharmacotherapy is still insufficient in the disease management. Transcatheter aortic valve implantation is recommended in selected groups of patients and provides optimal short and long-term outcomes.

Racial and ethnic disparities in aortic stenosis prevalence, management, and outcomes of treatment have been postulated. Data on discrepancies in aortic stenosis characteristics in patients qualified for transcatheter aortic valve implantation across populations are lacking.

The current project will conduct the analysis in populations of patients with aortic stenosis qualified for transcatheter aortic valve implantation from different countries to reveal potential disparities in clinical characteristics and in requirements for variations in prostheses sizes.

This is a retrospective, multicentre, observational registry of patients with severe aortic stenosis qualified for transcatheter aortic valve implantation.

Inclusion criteria - each site will include consecutive 100 patients who underwent transcatheter aortic valve implantation between January and June 2025.

Exclusion criteria - active infection (chronic inflammatory disease or neoplasm is not an exclusion criterion, however, will be considered in the laboratory analysis)

Data concerning

* patients' demographics,
* clinical characteristics
* results of aortic root and aorta analyses by computed tomography
* echocardiography results
* results of common laboratory tests (blood morphology, inflammatory ratios of neutrophils, monocytes and platelets to lymphocytes, glomerular filtration rate, N-terminal prohormone of brain natriuretic peptide) obtained during the routine care in the pre-procedural period will be collected at each site.

Simple procedural results (inc. prosthesis type and size) and outcomes (survival, bleeding, vascular complications, and acute kidney injury) will be recorded.

Collected data will be compared between study populations.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis qualified for TAVI

Exclusion Criteria:

* Active infection (chronic inflammatory disease or neoplasm is not an exclusion criterion, however, will be considered in the laboratory analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients qualified for TAVI will be included in the analysis and compared in subpopulations.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Aortic annulus diameter | Baseline
  Aortic annulus diameter in milimeters based on CT image
Aortic annulus area | Baseline
  Aortic annulus area in squared milimeters based on CT image
Aortic annulus perimeter | Baseline
  Aortic annulus perimeter in milimeters based on CT image
Ilio-femoral artery diameter | Baseline
  Ilio-femoral artery diameter in milimeter based on CT image
Neutrophils measured using whole blood count | Baseline
  This measurement is used to compute ratio of cell types using whole blood count
Monocytes measured in whole blood count | Baseline
  Number of monocytes identified in blood sample using automatic whole blood count. It is used to compute cell type ratio.
Lymphocytes measured using whole blood count | Baseline
  This measurement is used to compute ratio of cell types using whole blood count

CONTACTS AND LOCATIONS:
Overall Officials: Anna Olasinska-Wisniewska, Principal Investigator — Poznan University of Medical Sciences
Locations (5):
- San Bortolo's Hospital, Division of Cardiac Surgery and Division of Cardiology, Vicenza, Italy, Vicenza, Italy
- Poznan University of Medical Sciences, Poznan, Poland
- Institute for Cardiovascular Diseases of Vojvodina, Serbia University of Novi Sad, Novi Sad, Serbia
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand, Bangkok, Thailand
- Ankara Bilkent City Hospital, Ankara, Türkiye, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hakgor A, Dursun A, Kahraman BC, Yazar A, Savur U, Akhundova A, Olgun FE, Arman ME, Boztosun B. Prognostic impact of main pulmonary artery to ascending aorta diameter ratio in patients with severe aortic stenosis underwent transcatheter aortic valve implantation. Catheter Cardiovasc Interv. 2024 Apr;103(5):782-791. doi: 10.1002/ccd.31000. Epub 2024 Feb 28. PMID 38415894
- [Background] Yang Y, Richter R, Halfmann MC, Graafen D, Hell M, Vecsey-Nagy M, Laux G, Kavermann L, Jorg T, Geyer M, Varga-Szemes A, Emrich T. Prospective ECG-gated High-Pitch Photon-Counting CT Angiography: Evaluation of measurement accuracy for aortic annulus sizing in TAVR planning. Eur J Radiol. 2024 Sep;178:111604. doi: 10.1016/j.ejrad.2024.111604. Epub 2024 Jul 6. PMID 38996738
- [Background] Schafer M, Glotzbach JP, Sharma V, Tandar A, Welt FG, L Goodwin M, Smego D, Selzman CH, Pereira SJ. Aortic shape and diameter variations are predictive of short-term complications in transcatheter aortic valve replacement. Int J Cardiovasc Imaging. 2025 May;41(5):955-965. doi: 10.1007/s10554-025-03381-2. Epub 2025 Mar 29. PMID 40156693